CLINICAL TRIAL: NCT07118631
Title: Clinical Study on Emergency Treatment of Cerebral Arteriovenous Malformation Bleeding and Continuous Improvement of Medical Quality Based on Neurosurgery Hybrid Surgery Platform
Brief Title: Clinical Study on Emergency Treatment of Cerebral Arteriovenous Malformation Bleeding
Status: Recruiting | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BRWEP2024W022040104; BRWEP2024W022040104 (Other Grant/Funding Number: Beijing Municipal Health Commission)
Record Dates: First submitted 2025-07-30; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-07

CONDITIONS: Arteriovenous Malformation; Bleeding
Keywords: Cerebral hemorrhage; cerebral arteriovenous malformation; hybrid surgery; functional prognosis; quality improvement system
MeSH Terms: conditions — Arteriovenous Malformations; Hemorrhage; Cerebral Hemorrhage; Intracranial Arteriovenous Malformations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hybrid surgery cohort: After patients were enrolled, they were admitted to the hybrid operating room for DSA to confirm the diagnosis. If the patient meets the surgical indications, one-stop treatment with composite surgery will be performed. During the operation, the treatment plan is determined based on the characteristics of the malformation group, including simple embolization, partial embolization, auxiliary embolization for arteriovenous malformation resection, and the target area and proportion of embolization. For those who need craniotomy, the hematoma is removed during the operation and the brain arteriovenous malformation is removed under a microscope. Intraoperative ultrasound assists in locating the location, boundaries and residue of the malformation. Head DSA was reviewed immediately after surgery. Further clarify whether the lesions are completely removed. If the lesion remains, immediate surgical treatment and subsequent DSA review will be perfor

SUMMARY:
Cerebral arteriovenous malformation (AVM) is the leading cause of brain hemorrhage in young adults, characterized by sudden onset and rapid progression. The hybrid neurosurgical operating room is a diagnostic and therapeutic platform that integrates neurointervention and microneurosurgery, offering advantages such as one-stop rapid treatment and multimodal therapeutic approaches.

This study aims to focus on patients with acute cerebral AVM-related hemorrhage through a multicenter, prospective, registry-based research approach. In the hybrid neurosurgical operating room, emergency cerebral angiography, neurointerventional embolization, microsurgical resection of the vascular malformation, or minimally invasive hematoma evacuation will be performed to explore the indications and advantages of the hybrid neurosurgical operating platform in emergency AVM hemorrhage management. The study seeks to establish standardized diagnostic and treatment protocols and operational workflows for emergency AVM hemorrhage management in the hybrid operating room. Through continuous quality improvement, the study aims to further reduce patient morbidity and mortality.

This research will not only enhance the diagnostic and therapeutic level of cerebral AVM-related hemorrhage and improve patient outcomes but also effectively reduce medical costs and societal burdens.

ELIGIBILITY:
Inclusion Criteria:

* Head CT confirmed cerebral hemorrhage, with indications for emergency surgery
* Head CTA suggested that the responsible lesion may be cerebral arteriovenous malformation
* Spetzler-Martin classification 1 to 4; Cerebral arteriovenous malformation Spetzler-Martin classification is as follows: ① Nidus size: small (<3 cm) is scored as 1 point, medium (3 cm~6 cm) is scored as 2 points, and large (≥6 cm) is scored as 3 points; ② Adjacent brain functional areas: 0 points for non-functional areas, 1 point for functional areas; ③ Drainage veins: 0 points for superficial veins, 1 point for deep veins);
* Aged 18 to 70 years old, with systemic conditions that can tolerate surgery;
* Agree to surgical treatment and sign an informed consent form.

Exclusion Criteria:

* Consciousness disorder due to serious underlying diseases
* Patients or family members who refuse surgery
* Perinatal and pregnancy patients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with mergency cerebral arteriovenous malformation bleeding
Sampling Method: Probability Sample
Enrollment: 162 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Neurological outcomes | 2 weeks, 3 months, 6 months after surgery
  modified rankin scale (mRS), The scale runs from 0-6. Higher scores mean a worse outcome

SECONDARY OUTCOMES:
surgical information | pre-surgery, during the surgery, perioperatively immediately after the surgery
Complications | 2 weeks, 3 months, 6 months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No